CLINICAL TRIAL: NCT05007834
Title: Impact of Metabolic Status and Circadian Rhythms on Post-chemotherapy Ovarian Recovery in Women Treated for Breast Cancer
Brief Title: Metabolism, Circadian Rhythms and Ovarian Function
Acronym: METAB-OV
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_16; 2021-A00461-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-05-20; First posted 2021-08-16 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Chemotherapy-Induced Amenorrhea
Keywords: Ovarian recovery; Metabolism; Muscular mass; Adipose tissue; Chronotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chemotherapy for cancer, due to its gonadotoxicity, can lead to impaired female fertility, resulting in the occurrence of transient or prolonged chemo-induced amenorrhea (CIA). According to recent data from the National Cancer Institute, 11.9% of women under the age of 40 diagnosed with cancer have been offered a fertility evaluation within five years of diagnosis. Predicting the risk and especially the duration of the CIA remains difficult. Known factors predicting a rapid return of menstruation are a young age at diagnosis, a low gonadotoxic treatment (absence of alkylating agents) and a high pre-chemotherapy blood level of AMH reflecting a large pool of growing follicles. A body mass index (BMI) ≥ 25 kg / m² could also be a positive predictor, but this remains debated.

The objective of this project is to assess the impact of metabolism and energy reserves, physical activity and the chronotype on the recovery of ovarian function in patients with breast cancer who have developed CIA

ELIGIBILITY:
Inclusion Criteria:

* Women with a chemotherapy-induced (CIA) amenorrhea who asked for post-cancer fertility follow-up at the University Hospital of Lille, France.
* Women between 25 to 35 years age at inclusion
* Chemotherapy protocol: FEC 100 (3 cycles) + docetaxel (3 cycles

Exclusion Criteria:

* Women without CIA
* Women who refuse to participate in the study
* Women older than 35 years at inclusion
* Women who received another chemotherapy protocol

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with a chemotherapy-induced (CIA) amenorrhea
Study Population: Women with a chemotherapy-induced (CIA) amenorrhea who asked for post-cancer fertility follow-up at the University Hospital of Lille, France.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of IL-6 levels at the end of chemotherapy | 1 year
  Study the association between the IL-6 blood levels (in pg/ml) at the end of chemotherapy and the menstrual period return state ( before or after 6 months)

SECONDARY OUTCOMES:
Correlation between blood metabolic markers (Leptin, Insulin, Ghrelin) and menstrual period return state | 1 year
  Leptin concentration in ng/ml; insulin concentration in mUI/L; ghrelin concentrations in pg/ml
Correlation between physical activity score at the end of chemotherapy and menstrual period return state | 1 year
  Physical activity score expressed in arbitrary units
Correlation between chronotype score at the end of chemotherapy and menstrual period return state | 1 year
  chronotype score expressed in arbitrary units
Correlation between the BMI at the end of chemotherapy and menstrual period return state | 1 year
  weight and height will be combined to report BMI in kg/m2
Correlation between Blood metabolic markers (Leptin, Insulin, Ghrelin) assessed at 3 months and menstrual period return state | 9 months
  Leptin concentration in ng/ml, Insulin concentration in mUI/L, Ghrelin concentration in pg/ml
Correlation between the Physical activity Score at 3 months and the menstrual period return state (between 3 to 12 months) | 9 months
  Physical activity score expressed in arbitrary units
Correlation between the BMI assessed at 3 months and the menstrual period return state (between 3 to 12 months) | 9 months
  weight and height assessed at 3 months will be combined to report BMI in kg/m2
Evolution of the blood concentration of insulin over the follow-up period (12 months) | 1 year
  insulin concentrations expressed in mUI/L
Correlation between the Chronotype Score at 3 months and the menstrual period return state (between 3 to 12 months) | 9 months
  chronotype score expressed in arbitrary units
Evolution of the blood concentration of Leptin over the follow-up period (12 months) | 1 year
  leptin concentrations expressed in ng/ml
Evolution of the blood concentration of Ghrelin over the follow-up period (12 months) | 1 year
  ghrelin concentrations expressed in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Pascal PIGNY, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Jeanne de Flandre Chu Lille, Lille, France